CLINICAL TRIAL: NCT01433731
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Escalating Phase 1b Study to Assess the Safety, Pharmacodynamics and Pharmacokinetics of SHP 141, A Histone Deacetylase Inhibitor, Administered Topically Up to 28 Days to Patients With Stage IA, IB or IIA Cutaneous T-Cell Lymphoma
Brief Title: Safety, Pharmacodynamics (PD), Pharmacokinetics (PK) Study of SHP141 in 1A, 1B, or 2A Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TetraLogic Pharmaceuticals (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other); Therapeutics, Inc. (Industry); Veristat, Inc. (Other); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHP-141-001
Record Dates: First submitted 2011-09-09; First posted 2011-09-14 (Estimated); Results first posted 2016-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-01

CONDITIONS: Lymphoma, T-Cell, Cutaneous
Keywords: CTCL; Cutaneous T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo for SHAPE (SHP-141) (Placebo Comparator): placebo for SHAPE (SHHP-141) topical gelled solution
  Interventions: Drug: placebo for SHAPE (SHP-141)
- SHAPE (SHP-141) 0.1%BID (Experimental): SHAPE (SHP-141) topical gelled solution at 0.1% concentration twice weekly
  Interventions: Drug: SHAPE (SHP-141) 0.1% BID
- SHAPE (SHP-141) 0.5% BID (Experimental): SHAPE (SHP-141) topical gelled solution at 0.5% concentration twice weekly
  Interventions: Drug: SHAPE (SHP-141) 0.5% BID
- SHAPE (SHP-141) 1.0% BID (Experimental): SHAPE (SHP-141) topical gelled solution at 1.0% concentration twice weekly
  Interventions: Drug: SHAPE (SHP-141) 1.0% BID

INTERVENTIONS:
Drug: placebo for SHAPE (SHP-141) — topical gelled solution
  Arms: placebo for SHAPE (SHP-141)
Drug: SHAPE (SHP-141) 0.1% BID — topical gelled solution
  Arms: SHAPE (SHP-141) 0.1%BID
Drug: SHAPE (SHP-141) 0.5% BID — topical gelled solution
  Arms: SHAPE (SHP-141) 0.5% BID
Drug: SHAPE (SHP-141) 1.0% BID — topical gelled solution
  Arms: SHAPE (SHP-141) 1.0% BID

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of topical SHP141 applied directly to skin lesions in patients with Stage IA, IB, or IIA Cutaneous T-cell Lymphoma. This study will also investigate the effect of SHP141 on skin lesions in patients with Stage IA, IB, or IIA CTCL.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed CTCL; a documented verifiable biopsy report is required.
* Documented clinical Stage IA, IB, or IIA CTCL.
* Skin lesion involvement of at least 3% of BSA accessible for topical application of study drug and biopsy.
* ECOG performance status of 0-2.

Exclusion Criteria:

* CTCL with histologic evidence of folliculotropic variant or large cell transformed CTCL.
* Severe pruritus requiring systemic or topical treatment.
* Palpable lymph node ≥1.5 cm in diameter (unless the lymph node has been biopsied and has been designated as Stage IA-IIA disease).
* Coexistent second malignancy or history of prior solid organ malignancy within previous 5 years (excluding basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix (CIN 3), papillary or follicular thyroid cancer that has been treated curatively, or prostate cancer that has been treated curatively).
* Any prior history of a hematologic malignancy (other than CTCL).
* History of or current major renal, hepatic, gastrointestinal, pulmonary, cardiovascular, genito-urinary or hematological disease, CNS disorders, infectious disease or coagulation disorders as determined by the Investigator.
* Evidence of active Hepatitis B or C or HIV.
* Circulating atypical cells >5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Guitart, MD, Principal Investigator — Northwestern University
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - Northwestern University Dept of Dermatology, Chicago, Illinois
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Gahanna, Ohio
  - MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- SHAPE (SHP-141) 0.1% BID: SHAPE (SHP-141): topical gelled solution at 0.1% concentration twice daily
- SHAPE (SHP-141) 0.5% BID: SHAPE (SHP-141): topical gelled solution at 0.5% concentration twice daily
- SHAPE (SHP-141) 1.0% BID: SHAPE (SHP-141): topical gelled solution at 1.0% concentration twice daily
Period: Overall Study
Arm/Group | Placebo for SHAPE (SHP-141) | SHAPE (SHP-141) 0.1% BID | SHAPE (SHP-141) 0.5% BID | SHAPE (SHP-141) 1.0% BID
Started | 3 | 5 | 5 | 5
Completed | 3 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo for SHAPE (SHP-141): placebo for SHAPE (SHP-141): topical gel
- Total: Total of all reporting groups
Arm/Group | Placebo for SHAPE (SHP-141) | SHAPE (SHP-141) 0.1% BID | SHAPE (SHP-141) 0.5% BID | SHAPE (SHP-141) 1.0% BID | Total
Number analyzed (Participants) | 3 | 5 | 5 | 5 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 4 | 3 | 12
  >=65 years | 2 | 1 | 1 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 1 | 6
  Male | 2 | 2 | 4 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 5 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete or Partial Response as Measured by Change in Lesion Severity Using CAILS (Composite Assessment of Index Lesion Severity)
Description: Response assessed by change in lesion severity using Composite Assessment of Index Lesion Severity (CAILS) Assessment Tool which measures clinical signs of CTCL by erythema; scaling; plaque elevation; hypo- or hyperpigmentation, each on a scale of 0-8; and lesion size (cm2), on a scale of 0 (no lesion; 0 cm2) to 18 (300 cm2). Up to five index lesions are each scored, and a subtotal CAILS score is provided for each index lesion. A total score is calculated by summing these subtotals. Response criteria measure the change in CAILS score from baseline to follow-up as follows: Complete Response (CR): 100% decrease in CAILS score; Partial Response (PR): 50% - 99% decrease in CAILS score; Stable Disease (SD): < 25% increase to < 50% decrease in CAILS score; Progressive Disease (PD) ≥ 25% increase in CAILS score.
Time Frame: Weekly through day 28 (days 1, 7, 14, 21, 28) and again day 42
Measure: Number; unit: percentage of participants
Groups:
- SHAPE (SHP-141): Histone deacetylase inhibitor
  SHAPE (SHP-141): topical gel
Arm/Group | SHAPE (SHP-141) | Placebo for SHAPE (SHP-141)
Number analyzed (Participants) | 15 | 3
percentage of participants | 27 | 0

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Placebo for SHAPE (SHP-141) | SHAPE (SHP-141) 0.1% BID | SHAPE (SHP-141) 0.5% BID | SHAPE (SHP-141) 1.0% BID
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/3 | 5/5 | 4/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo for SHAPE (SHP-141) (N=3) | SHAPE (SHP-141) 0.1% BID (N=5) | SHAPE (SHP-141) 0.5% BID (N=5) | SHAPE (SHP-141) 1.0% BID (N=5)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Incision site blister (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Applications site warmth (General disorders) | 0 | 0 | 1 | 0
Edema peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No